CLINICAL TRIAL: NCT06724653
Title: Tapering Heart Failure Medication in Patients with Heart Failure with Recovered Ejection Fraction; Open Label Prospective Random Trial
Acronym: HFrecEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 2024-09-039-002; 2024-09-039-002 (Other: Chungnam national university hospital IRB)
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure; Ejection Fraction; Recovery of Function
Keywords: heart failure with recovered ejection fraction; Tapering
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: randomly assignment to 3 groups ( drug tapering_RAS blocker, beta blocker, drug maintaining)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RAS blocker tapering arm (Active Comparator): RAS blocker tapering
  Interventions: Drug: RAS blocker tapering group; Drug: Beta blocker tapering out
- Beta blocker tapering arm (Active Comparator): Beta blocker tapering arm
  Interventions: Drug: RAS blocker tapering group; Drug: Beta blocker tapering out
- Control (Placebo Comparator): Drug maintain group
  Interventions: Drug: RAS blocker tapering group; Drug: Beta blocker tapering out

INTERVENTIONS:
Drug: RAS blocker tapering group — RAS blocker tapering out
Drug: Beta blocker tapering out — Beta blocker tapering out group

SUMMARY:
Study start date is on Nov 27th 2024.

A patient with an initial ejection fraction (EF) of less than 40%, whose follow-up shows an improvement to an EF of 50% or higher, along with the left ventricular end-diastolic diameter returning to the normal range and taking 3 more heart failure medication randomed to drug tapering group ( RAS blocker or beta blocker) or continuing medication group.

DETAILED DESCRIPTION:
Patients described above randomly assigned to drug tapering group and drug maintaining group.

Drug tapering group is 2 groups, which one is RAS blocker tapering group and others is beta blocker tapering group.

Drug tapering group is monitored ejection fraction, LV dimension and LV GLS by 1-3 month.

ELIGIBILITY:
Inclusion Criteria:

* initial echocardiogram ejection fraction less than 40%
* follow up echocardiogram ejection fraction over 50% and LVEDD index normal range
* NTprobnp criteria

  1. eGFR ≥60 ; less 440
  2. eGFR 45-59: less 980
  3. eGFR 30-44; less 1220
  4. eGFR < 30 : less 5300
  5. in HD; no criteria for NTproBNP
* on more than 3 heart failure medication ( RAS blocker, beta blocker, mineral corticoid receptor antagonist, SGLT 2 inhibitor)

Exclusion Criteria:

1. under age 18 year
2. uncontrolled BP ( over 150/90)
3. coronary revascularization within 6 months
4. significant valve disease
5. arrhythmia requiring rate control
6. CKD with albuminuria ( over 30mg/g)
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-06 (Estimated); Primary Completion 2026-11-26 (Estimated); Study Completion 2027-11-26 (Estimated)

PRIMARY OUTCOMES:
Heart failure relapse | From enrollment to the end of treatment at 18 months
  LVEF 10% drop, EF less than 50 %, LVIDd/BSA 10% increase, over 33mm/m^2

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months after the publication of results with no end date